CLINICAL TRIAL: NCT05363930
Title: Randomized Controlled Trial Comparing Diagnostic Yield for Small Bowel Endoscopy Between Novel Motorized Spiral and Single Balloon Enteroscopy in Suspected Crohn's Disease (the MOTOR-CD Trial)
Brief Title: The MOTOR-CD Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MCD 1; version:1.0
Record Dates: First submitted 2022-04-28; First posted 2022-05-06 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Crohn's Disease
Keywords: Device-assisted enteroscopy; Single balloon enteroscopy; Novel motorized spiral enteroscopy; total enteroscopy
MeSH Terms: conditions — Crohn Disease | interventions — Single-Balloon Enteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single balloon enteroscopy (Active Comparator): Patients with suspected Crohn's disease requiring small bowel enteroscopy based on clinical features, laboratory investigation and in cross-sectional imaging (computed tomography/magnetic resonance enterography or enteroclysis/ video capsule endoscopy
  Interventions: Device: Single balloon enteroscopy
- Novel Motorized Spiral Enteroscopy (Active Comparator): Patients with suspected Crohn's disease requiring small bowel enteroscopy based on clinical features, laboratory investigation and in cross-sectional imaging (computed tomography/magnetic resonance enterography or enteroclysis/ video capsule endoscopy
  Interventions: Device: Novel motorized spiral enteroscopy

INTERVENTIONS:
Device: Novel motorized spiral enteroscopy — Novel motorized spiral enteroscopy (Olympus Medical Systems Corporation, Tokyo, Japan) procedures would be performed under general anaesthesia with nasotracheal intubation under fluoroscopic guidance. Four litres of PEG was given to all patients with at least 8 hours of fasting prior to NMSE. Initially antegrade enteroscopy would be performed failing which retrograde enteroscopy would be done to reach the lesion. If the desired lesion is not reached via antegrade/retrograde route, hemoclips would be applied or tattooing would be done followed by enteroscopy from opposite direction on the same day under the same anesthesia using the same overtube. The time of procedure will be calculated from insertion of NMSE to its withdrawal. The depth of insertion would be measured by sequential withdrawal technique.
  Arms: Novel Motorized Spiral Enteroscopy
Device: Single balloon enteroscopy — Single balloon enteroscopy will be performed with single balloon video-enteroscope (Olympus Medical Systems, Tokyo, Japan) under monitored anaesthesia (deep sedation with propofol). Initially antegrade/retrograde enteroscopy would be performed based on pre-procedure localization failing which enteroscopy would be done from opposite route to reach the lesion. Hemoclips would be applied or tattooing would be done followed by enteroscopy from opposite direction on the same day under the same anaesthesia using the same overtube. Duration of procedure would be calculated from the time of introduction of the enteroscope to time of removal. The depth of insertion would be measured using the push and pull technique.
  Arms: Single balloon enteroscopy

SUMMARY:
Both single-balloon enteroscopy (SBE) and novel motorized spiral enteroscopy (NMSE) are effective techniques for small bowel endoscopy in suspected Crohn's disease (CD). Small bowel endoscopy is indicated for confirming diagnosis when CD is suspected based on clinical features along with cross-sectional small bowel imaging (computed tomography enterography/enteroclysis: CTE or magnetic resonance enterography/enteroclysis: MRE) or capsule endoscopy (CE). It not only helps in diagnosing CD, but it also helps in excluding CD, diagnosing alternate conditions and taking a surgical decision if a tight stricture is found. The pilot study done by the investigators in 177 suspected CD patients (37.2% female, 7-75 years) undergoing total 201 device assisted enteroscopy (DAE) showed that NMSE scores over SBE with regards to small bowel evaluation with complete small bowel coverage and shorter procedure time. The investigators aim to validate this findings by comparing technical performance and diagnostic yield between NMSE (Olympus Medical, Tokyo, Japan) and SBE (Olympus Medical Systems Corporation, Tokyo, Japan) for small bowel evaluation. Additionally the investigators plan to compare depth of insertion, total enteroscopy rates, procedure time, adverse event rates between the two modalities.

To date, no study has compared both modalities in suspected Crohn's disease (CD) requiring small bowel evaluation in a randomized manner. Hence the investigators intend to perform a randomized controlled study based on these preliminary finding with appropriate matching and parallel study design in larger numbers.

DETAILED DESCRIPTION:
Study design

Study population Consecutive patients with suspected Crohn's disease requiring small bowel endoscopy based on abnormal imaging or capsule endoscopy shall be recruited.

Study settings:

The proposed study would be conducted in a high volume tertiary GI centre (Asian Institute of Gastroenterology) performing nearly more than 500 SBE/NMSE procedures per year with an well established inflammatory bowel disease (IBD) registry with more than 7000 IBD patients under follow up.

The study is approved by the institutional review boards and ethics committee. Written informed consent would be taken from each participants and the study would conform to the 1975 Declaration of Helsinki ethical guidelines.

Data collection A survey administration software (google forms) would be used to collect the participant data [age, sex, comorbidities, clinical features, smoking status, history of intestinal resection, type of DAE, indication of DAE, CT/MRE location and characteristic of lesions, capsule endoscopy findings, depth of insertion, time taken for the procedure, total enteroscopy rates, enteroscopy finding details, cause of failure if any, DAE findings, histopathology details, impact on management, adverse events, hospital stay and any therapeutic procedure performed e.g. endoscopic balloon dilation (EBD) with details]. Follow-up details for newly diagnosed CD cases would be collected via physical visit or telephonic communication.

Technique and instruments Single balloon enteroscopy: All SBE procedures will be performed with single balloon video-enteroscope (Olympus Medical Systems, Tokyo, Japan) under monitored anaesthesia (deep sedation with propofol). Initially antegrade/retrograde enteroscopy would be performed based on anticipated location in CT failing which enteroscopy would be done from opposite route to reach the lesion. If the desired lesion is not reached via antegrade/retrograde route, hemoclips would be applied or tattooing would be done followed by enteroscopy from opposite direction on the same day under the same anaesthesia using the same overtube. Fluoroscopy would be used in select cases with anticipated therapeutic procedure. All the procedures were done after minimum of 8 hours of fasting and bowel preparation was given with 4 litres of polyethylene glycol (PEG) for all. Duration of procedure would be calculated from the time of introduction of the enteroscope to time of removal. The depth of insertion would be measured using the push and pull technique. If the desired lesion is not reached by a single route and was deemed possible to reach by the other route, the area of maximal insertion shall be marked by India ink tattooing or hemoclip application followed by completion of bidirectional enteroscopy on the same or next working day.

Novel motorized spiral enteroscopy: All the NMSE (Olympus Medical Systems Corporation, Tokyo, Japan) procedures would be performed under general anaesthesia with nasotracheal intubation under fluoroscopic guidance. Four litres of PEG was given to all patients with at least 8 hours of fasting prior to NMSE. Initially antegrade enteroscopy would be performed failing which retrograde enteroscopy would be done to reach the lesion. If the desired lesion is not reached via antegrade route, hemoclips would be applied or tattooing would be done followed by retrograde enteroscopy on the same day under the same anesthesia using the same overtube. The time of procedure will be calculated from insertion of NMSE to its withdrawal. The depth of insertion would be measured by sequential withdrawal technique as described earlier.

All the enteroscopy procedures were performed by four small bowel endoscopists all of whom have performed at least 200 deep enteroscopy. At least 8 biopsies were taken from area of interest during DAE and sent for histopathological analysis. In selected cases, additional samples were sent for detection of tubercular bacilli using mycobacterium tuberculosis (MTB)-polymerase chain reaction (PCR) if clinically tuberculosis was considered as differential diagnosis. Histopathological findings were recorded under the following headings for diagnosing CD: chronic inflammation, architectural distortion and presence of granulomas.

Definitions:

Technical success shall be defined as enteroscope introduction beyond duodenojejunal (DJ) flexure or ileocecal valve via antegrade and retrograde route respectively. The diagnostic yield with DAE shall be defined as the percentage of procedures which confirmed/excluded lesions found on prior cross-sectional imaging (CTE/MRE) or found new/alternate diagnosis explaining the clinical condition. Depth of maximal insertion (DMI) will be defined as the point beyond which DAE advancement was not feasible. Major adverse events are perforation, pancreatitis, bleeding requiring transfusion or procedure related hospitalization. Minor adverse events are superficial mucosal injury, self limiting sore throat/nausea/vomiting, minor bleeding (without need for blood transfusion) or pain abdomen (not requiring hospital admission). Total enteroscopy will be defined as examination of small bowel from DJ flexure to ileocecal valve. Total enteroscopy would be achieved by either uni-directional (antegrade or retrograde route) or bi-directional enteroscopy (using both antegrade and retrograde route). The histopathological diagnosis of CD will be confirmed if non-caseating micro-granulomas are found with either of both of the other two histological features (chronic inflammation and architectural distortion) and alternate diagnosis like small bowel tuberculosis is ruled out based on clinical, radiologic and other relevant findings. Presence of both chronic inflammation and architectural distortion, non-caseating granuloma/chronic inflammation/ architectural distortion alone will be considered suggestive of CD in the appropriate clinical settings.

Sample size

Based on the pilot study by the investigators, diagnostic yield for deep enteroscopy with NMSE and SBE (97.8% and 83.2% respectively, the estimated sample size is total 124 (62 in each group) keeping type 1 error as 0.05 and power as 80%.

Randomisation

Randomisation will be done based on web based randomisation services

Timeline: 2 years Recruitment of 124 suspected CD patients requiring small bowel evaluation over maximum 2 years.

Patient privacy An organised database for the purpose of this study will be formed based on google form with anonymised data set (i.e. name, address, and full post code will be removed, together with any other information which, in conjunction with other data held by or disclosed to the recipient, could identify the patient) which would be entered by clinical research assistant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected of known IBD requiring small bowel endoscopy
2. Ability to give a signed informed consent.
3. Age ≥18 years -65 years -

Exclusion Criteria:

1. Patient not fit for general anaesthesia
2. Pediatric Patients (<18 years)
3. Pregnant or lactating mother
4. Post operative cases
5. Not willing to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Comparison of technical success with NMSE and SBE per patient [%] | 2 years
  Percentage of participants in which anatomical region of interest is reached

SECONDARY OUTCOMES:
Comparison of diagnostic yield with NMSE and SBE per procedure [%] | 2 years
  Percentage of enteroscopy procedures in which Crohn's disease or other disease is diagnosed or ruled out
Comparison of procedure time with NMSE and SBE[minutes] | 2 years
  Time from enteroscope insertion to withdrawal
Comparison of depth of maximal insertion with NMSE and SBE [centimetres] | 2 years
  Maximum depth reached by NMSE/SBE from duodenojejunal flexure for antegrade and ileocecal valve for retrograde enteroscopy
Comparison of total enteroscopy rates with NMSE and SBE [percentage] | 2 years
  Percentage of cases in which total small bowel examination is performed
Comparison of adverse events with NMSE and SBE [percentage] | 2 years
  Major adverse events are perforation, pancreatitis, bleeding requiring transfusion or procedure related hospitalization. Minor adverse events are superficial mucosal injury, self limiting sore throat/nausea/vomiting, minor bleeding (without need for blood transfusion) or pain abdomen (not requiring hospital admission).

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

REFERENCES:
- [Derived] Pal P, Ramchandani M, Banerjee R, Viswakarma P, Singh AP, Reddy M, Rughwani H, Patel R, Sekaran A, Kanaganti S, Darisetty S, Nabi Z, Singh J, Gupta R, Lakhtakia S, Pradeep R, Venkat Rao G, Tandan M, Reddy DN. Technical performance and diagnostic yield of motorised spiral enteroscopy compared with single-balloon enteroscopy in suspected Crohn's disease: a randomised controlled, open-label study (the MOTOR-CD trial). Gut. 2023 Oct;72(10):1866-1874. doi: 10.1136/gutjnl-2023-329885. Epub 2023 May 17. PMID 37197904